CLINICAL TRIAL: NCT03119064
Title: BrUOG 329: Onivyde (Nanoliposomal Irinotecan) and Metronomic Temozolomide for Patients With Recurrent Glioblastoma: A Phase IB/IIA Brown University Oncology Research Group Study
Brief Title: BrUOG 329 Onivyde & Metronomic Temozolomide in Recurrent Glioblastoma
Acronym: 329
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of response to study therapy
Sponsor: Brown University (Other)
Collaborators: Merrimack Pharmaceuticals (Industry); Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BrUOG 329
Record Dates: First submitted 2017-04-06; First posted 2017-04-18 (Actual); Results first posted 2022-02-24 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Glioblastoma Multiforme; Glioblastoma; GBM
MeSH Terms: conditions — Glioblastoma | interventions — irinotecan sucrosofate; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose 1 (Experimental): Temozolomide: 50mg/m2/day until disease progression.
  Nanoliposomal irinotecan :
  Dose Level 1 50mg/m2 IV every 2 weeks
  Interventions: Drug: Nanoliposomal Irinotecan; Drug: Temozolomide
- Dose 2 (Experimental): Temozolomide: 50mg/m2/day until disease progression.
  Nanoliposomal irinotecan :
  Dose Level 2 70 mg/m2 IV every 2 weeks
  Interventions: Drug: Nanoliposomal Irinotecan; Drug: Temozolomide
- Dose 3 (Experimental): Temozolomide: 50mg/m2/day until disease progression.
  Nanoliposomal irinotecan :
  Dose Level 3 80mg/m2 IV every 2 weeks
  Interventions: Drug: Nanoliposomal Irinotecan; Drug: Temozolomide

INTERVENTIONS:
Drug: Nanoliposomal Irinotecan — Three patients will be accrued to level 1. If no dose limiting toxicities are observed following completion of 4 weeks (2 cycles) of treatment then accrual to dose level 2 will proceed (patients must be evaluated prior to their cycle 3 treatment and this will be used to confirm DLTs). If a DLT is observed in one of the first 3 patients in a dose level, then accrual for that level will be expanded to 6 patients. Accrual will continue in this way until the MTD of nanoliposomal irinotecan with temozolomide 50mg/m2/day is determined. Two or more instances of DLT in a cohort of 6 patients will result in the preceding dose level being defined as the MTD. If two or more instances of DLT in a cohort of 6 patients occurs in dose level 1 then dose level -1 of nanoliposomal irinotecan will be investigated. After determination of the MTD, the final cohort will be expanded so that a total of 25 patients are treated on study. The final cohort will be treated at the MTD.
  Other Names: Onivyde
Drug: Temozolomide — Three patients will be accrued to level 1. If no dose limiting toxicities are observed following completion of 4 weeks (2 cycles) of treatment then accrual to dose level 2 will proceed (patients must be evaluated prior to their cycle 3 treatment and this will be used to confirm DLTs). If a DLT is observed in one of the first 3 patients in a dose level, then accrual for that level will be expanded to 6 patients. Accrual will continue in this way until the MTD of nanoliposomal irinotecan with temozolomide 50mg/m2/day is determined. Two or more instances of DLT in a cohort of 6 patients will result in the preceding dose level being defined as the MTD. If two or more instances of DLT in a cohort of 6 patients occurs in dose level 1 then dose level -1 of nanoliposomal irinotecan will be investigated. After determination of the MTD, the final cohort will be expanded so that a total of 25 patients are treated on study. The final cohort will be treated at the MTD.
  Other Names: TMZ

SUMMARY:
New treatments are greatly needed for patients with recurrent glioblastoma. Metronomic temozolomide is a standard treatment option but has, at best, modest activity. The nanoliposomal irinotecan may be much more active than the parent compound irinotecan since nanoliposomal irinotecan's ability to cross the blood brain barrier is improved. This phase I study will establish the MTD of the combination of nanoliposomal irinotecan in combination with temozolomide safety and preliminary clinical efficacy of the combination of nanoliposomal irinotecan and metronomic temozolomide.

DETAILED DESCRIPTION:
1.1 Primary Objective 1.1.1. To evaluate the maximum tolerated dose of nanoliposomal irinotecan with continuous low-dose temozolomide for patients with recurrent glioblastoma.

1.1.2 To assess the preliminary response rate and progression free survival of nanaliposomal irinotecan with continuous low-dose temozolomide in patients with recurrent glioblastoma.

1.2 Secondary Objectives 1.2.1 To evaluate the safety of nanoliposomal irinotecan with continuous low-dose temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma multiforme (gliosarcoma also eligible), Pathology report to be sent to BrUOG.
* Progression or recurrence after at least one line of therapy. Patient must have received temozolomide and radiation but it is not required that they were given concurrently.
* Age >18 years
* Karnofsky performance score > 60
* Life expectancy >12 weeks as noted by treating investigator
* Laboratory results requirements

  * Absolute neutrophil count (ANC) ≥ 1500/mm3.
  * Platelets (Plt) ≥ 100,000/mm3
  * Hemoglobin (Hgb) ≥ 9.0 g/dL
  * Total bilirubin < 1x ULN
  * Albumin levels ≥ 3.0 g/dL
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x ULN
  * Serum creatinine ≤ 1.5 x ULN
* Not pregnant and not nursing. Women of child bearing potential must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days prior to Day 1 of treatment. Post-menopausal women (surgical menopause or lack of menses >12 months) do not need to have a pregnancy test, please document status.
* Confirmation of informed consent.
* Men and women of childbearing potential enrolled in this study must agree to use adequate barrier birth control measures during the course of the study and for at least 2 months after the last treatment on study.
* Recovered (< grade 1) from clinically significant effects of any prior surgery, radiotherapy or other anti-neoplastic therapy, except alopecia or hematological laboratory values
* Stable corticosteroid dose at least 7 days prior to day 1
* Patients must have assessable (measurable) disease at baseline by brain MRI. Must be contrast enhancing. The tumor size will be measured in millimeters and is the largest cross-sectional area using perpendicular measurements of contrast enhancing abnormality.
* Patient must be able to tolerate brain MRI with contrast

Exclusion Criteria:

* Non-GBM primary invasive malignant neoplasm that is considered by treating investigator to likely cause death in the next 5 years.
* Radiation therapy or cytotoxic chemotherapy or biologics or immunotherapy within previous three weeks from day 1 of drug (no anticancer treatment of any kind within 3 weeks of day 1 of drug- steroids are acceptable if stable dose per 3.1.11).
* Patients not to be receiving any cancer therapy or investigational anti-cancer drug.
* Evidence of an active infection requiring intravenous antibiotic therapy
* Any medical condition that in the opinion of the Investigator may interfere with a subject's participation in or compliance with the study. Must receive confirmation in writing from treating MD.
* Pregnant or breast feeding; females of child-bearing potential must test negative for pregnancy at the time of enrollment based on serum pregnancy test.
* Unwillingness or inability to follow the procedures required in the protocol, site to have documentation to confirm at time of registration that this is not the case.
* Patient with a history of Gilbert's disease or known UGT1A1*28 allele. (Assessment for the UGT1A1*28 allele is not required for protocol entry.) Documentation required at time of study entry by treating MD.
* myocardial infarction, unstable angina pectoris, stroke within 6 months of study registration.
* NYHA Class III or IV congestive heart failure
* Known hypersensitivity to any of the components of nanoliposomal irinotecan , other liposomal products, or temozolomide. Must be documented by treating MD.
* Investigational anticancer therapy administered within 4 weeks of day 1, or within a time interval less than at least 5 half lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study. Site must submit all prior investigational agents with last dose administered and half-life for BrUOG review.
* Live vaccines within 30 days prior to the first dose of trial treatment and while participating in the trial. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, BCG, and typhoid (oral) vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines and are not allowed. All recent vaccines (within 30 days) to be listed on conmed log and submitted to BrUOG.
* Use of strong CYP3A4 inducers is not allowed and patients must be off any of these exclusionary products for > 2 weeks from day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Safran, MD, Study Chair — BrUOG Study Chair
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elinzano H, Toms S, Robison J, Mohler A, Carcieri A, Cielo D, Donnelly J, Disano D, Vatketich J, Baekey J, Sturtevant A, MacKinnon K, Wood R, Safran H. Nanoliposomal Irinotecan and Metronomic Temozolomide for Patients With Recurrent Glioblastoma: BrUOG329, A Phase I Brown University Oncology Research Group Trial. Am J Clin Oncol. 2021 Feb 1;44(2):49-52. doi: 10.1097/COC.0000000000000780. PMID 33284237

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose 1 | Dose 2 | Dose 3
Started | 9 | 3 | 0
Completed | 9 | 3 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose 1 | Dose 2 | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 9
  >=65 years | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: years] | 54 [39 to 70] | 64 [58 to 71] | 56 [39 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 8 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 8 | 3 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Determination of Maximum Tolerated Dose (MTD)
Description: To evaluate the maximum tolerated dose of nanoliposomal irinotecan with continuous low-dose temozolomide for patients with recurrent glioblastoma.
Time Frame: Every two weeks for 4 weeks
Measure: Number; unit: mg/m^2
Groups:
- All Participants: Temozolomide: until disease progression.
  Nanoliposomal irinotecan : IV every 2 weeks
Arm/Group | All Participants
Number analyzed (Participants) | 12
mg/m^2 | 50

2. Primary Outcome: Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR."
Time Frame: Every 2 months on study treatment then very 3 months once treatment has stopped, until progression of disease up to 2 years.
Measure: Number; unit: participants
Arm/Group | Dose 1 | Dose 2
Number analyzed (Participants) | 9 | 3
participants
  Partial Response | 1 | 1
  Progressive Disease | 8 | 2

3. Primary Outcome: Survival Status of Participants Treated With Nanaliposomal Irinotecan With Continuous Low-dose Temozolomide in Patients With Recurrent Glioblastoma.
Time Frame: Collected every 3 months once treatment has stopped, until progression of disease, up to 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose 1 | Dose 2
Number analyzed (Participants) | 9 | 3
Participants
  Deceased | 8 | 2
  Alive | 1 | 1

4. Secondary Outcome: Toxicities
Description: Treatment emergent toxicities of nanoliposomal irinotecan with continuous low-dose temozolomide using CTCAE version 4.03, grades 2 through 4
Time Frame: Baseline through 30 days post off study treatment
Measure: Number; unit: events
Arm/Group | Dose 1 | Dose 2
Number analyzed (Participants) | 9 | 3
events
  Neutropenia | 0 | 1
  ALT/AST | 2 | 1
  Hypokalemia | 1 | 1
  Hypophosphatemia | 1 | 0
  Nausea | 1 | 2
  Fatigue | 2 | 2
  Diarrhea | 0 | 2
  Anorexia | 0 | 2
  Dehydration | 0 | 2
  Urticaria | 1 | 0

ADVERSE EVENTS:
Time Frame: From time of study consent until 30 days after the last dose of study treatment, an average of 6 months.
Arm/Group | Dose 1 | Dose 2
All-Cause Mortality (participants affected / at risk) | 8/9 | 2/3
Serious Adverse Events (participants affected / at risk) | 4/9 | 3/3
Other Adverse Events (participants affected / at risk) | 9/9 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 (N=9) | Dose 2 (N=3)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebral edema (Nervous system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0 — Right femoral neck
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Acute pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Thromboembolic event (Vascular disorders) | 2 | 0
Craniotomy (Surgical and medical procedures) | 3 | 0
Muscle weakness right-sided (Nervous system disorders) | 0 | 1
C.diff (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose 1 (N=9) | Dose 2 (N=3)
Agitation (Psychiatric disorders) | 1 | 0
ALT increased (Investigations) | 3 | 1
Anxiety (Psychiatric disorders) | 1 | 0
AST increased (Investigations) | 2 | 1
Cognitive distrubance (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 2
Dizziness (Nervous system disorders) | 2 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Edema limbs (General disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 2
Fatigue (General disorders) | 3 | 2
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
GERD (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 2
Hypertension (Vascular disorders) | 2 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Pain (General disorders) | 2 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 | 0
Platelet count decreased (Investigations) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Seizure (Nervous system disorders) | 2 | 0
Weight loss (Investigations) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-12-08): https://cdn.clinicaltrials.gov/large-docs/64/NCT03119064/Prot_SAP_ICF_000.pdf